CLINICAL TRIAL: NCT02718859
Title: Study of the Combined Therapy of Irreversible Electroporation（IRE） and Nature Killer (NK) Cells for Advanced Pancreatic Cancer
Brief Title: Combination of Irreversible Electroporation and NK Immunotherapy for Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Shenzhen Hank Bioengineering Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK-pancre
Record Dates: First submitted 2016-03-09; First posted 2016-03-24 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-03

CONDITIONS: Pancreatic Cancer
Keywords: advanced pancreatic cancer; nature killer cell; irreversible electroporation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- irreversible electroporation (IRE) (Active Comparator): Advanced pancreatic cancer patients received only irreversible electroporation (IRE) without immunotherapy
  Interventions: Procedure: irreversible electroporation (IRE )
- IRE & NK cells (Experimental): Advanced pancreatic cancer patients received both irreversible electroporation (IRE ) and immunotherapy of nature killer(NK) cells
  Interventions: Biological: NK cells; Procedure: irreversible electroporation (IRE )

INTERVENTIONS:
Biological: NK cells — The pancreatic cancer patients will receive nature killer(NK) cells infusions,qd
  Arms: IRE & NK cells
Procedure: irreversible electroporation (IRE ) — The pancreatic cancer patients will receive the therapy of irreversible electroporation (IRE )

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the combined therapy using irreversible electroporation（IRE）and nature killer(NK) cells for advanced pancreatic cancer.

DETAILED DESCRIPTION:
By enrolling patients with pancreatic cancer adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of the combined therapy using irreversible electroporation（IRE）and nature killer（NK） cells for advanced pancreatic cancer.

The efficacy will be evaluated according to relief degree,progress free survival(PFS) and overall survival(OS).

The safety will be evaluated by statistics of adverse reaction

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-80
2. Diagnosis：advanced and active pancreatic cancer
3. The tumour is measurable
4. Eastern Cooperative Oncology Group(ECOG) score：0~2；3 but has no relationship with tumour
5. Vital organ function is normal:

   total bilirubin(TB) <68μmol/L aspartate aminotransferase(AST)<90 IU/L Cre<353μmol/L white blood cell count(WBC)<9×10^9/L,when WBC is close to or even greater than 9×10^9/L，the recommended dose should be halved platelet count(PLT)>80×10^9/L Red blood cell specific volume(HCT)>0.20 Non severe viral or bacterial infection
6. Non pregnant and lactating patients
7. Non allergic reactions to biological products
8. Informed and consent

Exclusion Criteria:

1. Patients with cardiac pacemaker
2. Patients with severe cardiac and pulmonary dysfunction
3. Patients that the researchers do not think fit into the group,including patients failed in compliance assessment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Relief degree | 1 year
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors（RECIST）

SECONDARY OUTCOMES:
Progress free survival（PFS） | 1 year
Overall survival（OS） | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, PhD, Study Chair — Fuda Cancer Hospital
Locations (1):
- Central laboratory in Fuda cancer hospital, Guangzhou, Guangdong, China